CLINICAL TRIAL: NCT00186602
Title: Does a Peer Navigator Improve Quality of Life at Diagnosis?
Brief Title: Does a Peer Navigator Improve Quality of Life at Diagnosis for Women With Breast Cancer?
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: California Breast Cancer Research Program (Other); Genentech, Inc. (Industry); Amgen (Industry); Johnson & Johnson (Industry); Google LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: 7BB-2400; 12382 (Other: Stanford-IRB)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2005-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Behavioral: Peer counseling

SUMMARY:
Women indicate the greatest needs for counseling at the time of initial diagnosis for primary breast cancer. The time of initial diagnosis is also often the time of greatest need for information for women and their families. However, this is the time when a woman, overwhelmed by shock and trauma, is least likely to absorb information provided or seek new sources of information. An informed peer navigator with carefully trained communication skills can judge the level of information to disclose and pace that information in a way that can be easily absorbed and understood. She will also provide support. WomenCARE, a well-established Santa Cruz agency providing free support services for women with cancer, and the Psychosocial Treatment Lab at Stanford therefore ask whether women newly diagnosed with breast cancer will improve their quality of life by participating in a peer navigator program. WomenCARE's peer navigators provide emotional support, good listening skills, and information on resources for women just diagnosed with breast cancer. Having a peer counselor while a woman goes through treatment may reduce the magnitude of distress or shorten its time course. It may also reduce distress in family members, and improve relationships with medical personnel.

This study is designed to evaluate the effectiveness of a peer navigator program where a woman newly diagnosed with breast cancer is carefully matched for 3 to 6 months after diagnosis with a trained volunteer who is herself a breast cancer survivor. Navigators and Sojourners (newly diagnosed women) are matched on things that are important to them. Women often want to be matched on the type of surgery or treatment they have received. We assign half of the women (by a process similar to a coin toss) to our peer navigator program and half to a group that receives standard medical care but no peer navigator. In this way we can compare the groups to see whether those matched with a peer navigator have better quality of life over the 3 to 6 month period. All women who join our study, regardless of the group to which they are assigned, get an extra consultation with a nurse specialist at a local hospital. In this consultation, the nurse reviews the cancer resources available to the woman in Santa Cruz County. This meeting is tailored to the woman's individual diagnosis and situation.

ELIGIBILITY:
Inclusion Criteria:

women within 2 months of diagnosis of breast cancer can read English within the catchment area of Watsonville and Santa Cruz California -

Exclusion Criteria:

women who have previously had a peer navigator intervention women who have a chronic history of hospitalization for psychiatric reason

-

Ages: 20 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2000-07-01 (Actual); Primary Completion 2006-11-30 (Actual); Study Completion 2006-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, M.D., Principal Investigator — Stanford University; Caroline Bliss-Isberg, Ph.D., Principal Investigator — Cabrillo College; Janine Giese-Davis, Ph.D., Study Director — Stanford University
Locations (1):
- WomenCARE, Santa Cruz, California, United States